CLINICAL TRIAL: NCT06329986
Title: A Randomized, Crossover Controlled Trial of the Effect of TAMER Lenses Versus Single Vision Lenses on Myopic Progression in Myopic Children
Brief Title: Crossover RCT of TAMER Lenses in Myopia Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SEDPTC20240109
Record Dates: First submitted 2024-02-01; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-01

CONDITIONS: Myopia; Progressive
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): TAMER lenses are used first for 6 months, followed by SV lenses for 6 months.
  Interventions: Device: TAMER Lens Spectacle; Device: SV lenses
- Group B (Experimental): SV lenses are used first for 6 months, followed by TAMER lenses for 6 months.
  Interventions: Device: TAMER Lens Spectacle; Device: SV lenses

INTERVENTIONS:
Device: TAMER Lens Spectacle — Regular daily wear of TAMER lens spectacle
Device: SV lenses — SV lenses

SUMMARY:
This study is a prospective, randomized, crossover clinical trial with a planned proposed enrollment of 120 Chinese male and female subjects aged 6-12 years without systemic or ocular diseases to follow up their cycloplegic equivalent spherical lens power and other relevant indices in order to determine the role of TAMER lenses in myopia control as compared to singlie vision lenses.

ELIGIBILITY:
Inclusion Criteria:

* Race: Chinese children and adolescents.
* Age 6-12 years, gender unrestricted.
* Cycloplegic refraction SER: -0.75DS~-5.0DS in both eyes.
* Best corrected visual acuity of both eyes reaches 0.8 (0.00 logMAR).
* Cylinder power and astigmatism are no more than 1.5D.
* During the study period, willing to wear glasses provided by the researcher only and without additional interventions.
* Willing to be randomly assigned.
* Able to sign an informed consent form with the accompaniment and understanding of parents or guardians.

Exclusion Criteria:

* Allergic or intolerant to medications used for cycloplegia.
* Received any nearsightedness treatment such as atropine, rigid gas permeable contact lens, bifocal/progressive lens, red light therapy, or acupuncture within half a year before the study.
* Diagnosed with any eye disease other than nearsightedness, including strabismus, corneal diseases, conjunctival or eyelid damage or other conditions (such as keratoconus, herpes simplex keratitis, etc.).
* History of eye surgery (including strabismus correction surgery).
* Eye or systemic diseases that might be associated with nearsightedness or its progression, such as Marfan syndrome, retinopathy of prematurity, diabetes, etc.
* Anatomical or dermatological factors that may interfere with the wearing of spectacle frames.
* Other reasons that the researcher deems inappropriate for the participant to be included in the study, such as excessively high expectations for the effectiveness of defocus lenses, or plans to use other nearsightedness intervention strategies simultaneously with the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Spherical Equivalent change | 6 months
  cycloplegic SE change

SECONDARY OUTCOMES:
Axial Length change | 6 months
Spherical Equivalent change | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality, China